CLINICAL TRIAL: NCT03969888
Title: A Phase 2 Study of ABBV-3067 Alone and in Combination With ABBV-2222 in Cystic Fibrosis Subjects Who Are Homozygous for the F508del Mutation
Brief Title: A Phase 2 Study of ABBV-3067 Alone and in Combination With ABBV-2222
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M19-530; 2019-000750-63 (EudraCT Number)
Record Dates: First submitted 2019-05-30; First posted 2019-05-31 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; ABBV-3067; ABBV-2222, F508del Mutation
MeSH Terms: conditions — Cystic Fibrosis | interventions — GLPG2222

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- ABBV-3067 50 mg + Placebo for ABBV-2222 (Experimental): Participants received ABBV-3067 50 mg tablet orally once daily (QD) plus placebo matching ABBV-2222 capsule, orally QD for 28 days.
  Interventions: Drug: ABBV-3067; Drug: Placebo ABBV-2222
- ABBV-3067 150 mg + Placebo for ABBV-2222 (Experimental): Participants received ABBV-3067 150 mg tablet orally QD plus placebo matching ABBV-2222 capsule, orally QD for 28 days.
  Interventions: Drug: ABBV-3067; Drug: Placebo ABBV-2222
- ABBV-3067 150 mg + ABBV-2222 10 mg (Experimental): Participants received ABBV-3067 150 mg tablet orally QD plus ABBV-2222 10 mg capsule orally QD for 28 days.
  Interventions: Drug: ABBV-3067; Drug: ABBV-2222
- ABBV-3067 150 mg + ABBV-2222 30 mg (Experimental): Participants received ABBV-3067 150 mg tablet orally QD plus ABBV-2222 30 mg capsule orally QD for 28 days.
  Interventions: Drug: ABBV-3067; Drug: ABBV-2222
- ABBV-3067 150 mg + ABBV-2222 100 mg (Experimental): Participants received ABBV-3067 150 mg tablet orally QD plus ABBV-2222 100 mg capsule orally QD for 28 days.
  Interventions: Drug: ABBV-3067; Drug: ABBV-2222
- ABBV-3067 150 mg + ABBV-2222 200 mg (Experimental): Participants received ABBV-3067 150 mg tablet orally QD plus ABBV-2222 200 mg capsule, orally QD for 28 days.
  Interventions: Drug: ABBV-3067; Drug: ABBV-2222
- ABBV-3067 150 mg + ABBV-2222 300 mg (Experimental): Participants received ABBV-3067 150 mg tablet orally QD plus ABBV-2222 300 mg capsule, orally QD for 28 days.
  Interventions: Drug: ABBV-3067; Drug: ABBV-2222
- Placebo for ABBV-3067 + Placebo for ABBV-2222 (Placebo Comparator): Participants received placebo matching ABBV-3067 tablet orally QD plus placebo matching ABBV-2222 capsule, orally QD for 28 days.
  Interventions: Drug: Placebo ABBV-3067; Drug: Placebo ABBV-2222

INTERVENTIONS:
Drug: ABBV-3067 — Tablet taken orally.
  Arms: ABBV-3067 150 mg + ABBV-2222 10 mg; ABBV-3067 150 mg + ABBV-2222 100 mg; ABBV-3067 150 mg + ABBV-2222 200 mg; ABBV-3067 150 mg + ABBV-2222 30 mg; ABBV-3067 150 mg + ABBV-2222 300 mg; ABBV-3067 150 mg + Placebo for ABBV-2222; ABBV-3067 50 mg + Placebo for ABBV-2222
Drug: Placebo ABBV-3067 — Tablet taken orally.
  Arms: Placebo for ABBV-3067 + Placebo for ABBV-2222
Drug: ABBV-2222 — Capsule taken orally.
  Arms: ABBV-3067 150 mg + ABBV-2222 10 mg; ABBV-3067 150 mg + ABBV-2222 100 mg; ABBV-3067 150 mg + ABBV-2222 200 mg; ABBV-3067 150 mg + ABBV-2222 30 mg; ABBV-3067 150 mg + ABBV-2222 300 mg
Drug: Placebo ABBV-2222 — Capsule taken orally.
  Arms: ABBV-3067 150 mg + Placebo for ABBV-2222; ABBV-3067 50 mg + Placebo for ABBV-2222; Placebo for ABBV-3067 + Placebo for ABBV-2222

SUMMARY:
This study will evaluate the safety, tolerability, and efficacy of ABBV-3067 given alone and in combination with various doses of ABBV-2222 in adults with Cystic Fibrosis who are homozygous for the F508del mutation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of Cystic Fibrosis (CF) who are homozygous for the F508del CF transmembrane conductance regulator (CFTR) mutation
* Stable pulmonary status
* Lung function >= 40 and <= 90% of predicted normal for age, gender and height at Screening

Exclusion Criteria:

* History of solid organ or hematopoietic transplant
* Cirrhosis with portal hypertension
* Use of CFTR modulator therapy within 60 days prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (51):
- United States (10):
  - University of Arkansas /ID# 212541, Little Rock, Arkansas
  - Tampa General Hospital /ID# 212342, Tampa, Florida
  - University of Iowa Hospitals and Clinics /ID# 212351, Iowa City, Iowa
  - Univ Michigan Med Ctr /ID# 212657, Ann Arbor, Michigan
  - Cardinal Glennon Children's Hospital /ID# 212349, St Louis, Missouri
  - Washington University-School of Medicine /ID# 212352, St Louis, Missouri
  - Nationwide Children's Hospital /ID# 213158, Columbus, Ohio
  - Medical University of South Carolina /ID# 212187, Charleston, South Carolina
  - Vanderbilt University Medical Center /ID# 212353, Nashville, Tennessee
  - University of Utah /ID# 212350, Salt Lake City, Utah
- Belgium (5):
  - Uza /Id# 213412, Edegem, Antwerpen
  - Cliniques Universitaires de Bruxelles Hopital Erasme /ID# 213413, Brussels, Brussels Capital
  - UZ Brussel /ID# 212812, Jette, Brussels Capital
  - UZ Gent /ID# 213411, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 213050, Leuven, Vlaams-Brabant
- Canada (7):
  - University of Calgary /ID# 212555, Calgary, Alberta
  - St. Paul's Hospital /ID# 212554, Vancouver, British Columbia
  - QEII - Health Sciences Centre /ID# 212656, Halifax, Nova Scotia
  - Unity Health Toronto - St. Michael's Hospital /ID# 212552, Toronto, Ontario
  - CHUM - Centre hospitalier de l'Universite de Montréal /ID# 227815, Montreal, Quebec
  - McGill University Health Center Research Institute /ID# 212553, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec - Université L /ID# 212655, Québec, Quebec
- Czechia (2):
  - Fakultni Nemocnice Brno /ID# 213437, Brno
  - Fakultni Nemocnice v Motole /ID# 212966, Prague
- France (8):
  - Chu de Nice-Hopital L'Archet Ii /Id# 212862, Nice, Alpes-Maritimes
  - HCL - Hopital Lyon Sud /ID# 212899, Pierre-Bénite, Auvergne-Rhône-Alpes
  - CHU Bordeaux - Hopital Haut Leveque /ID# 212898, Pessac, Gironde
  - CHU Montpellier - Hôpital Saint Eloi /ID# 212856, Montpellier, Herault
  - AP-HP - Hopital Cochin /ID# 212864, Paris
  - CHU de Reims - Hôpital Maison Blanche /ID# 212910, Reims
  - Fondation ILDYS /ID# 212857, Roscoff
  - CHU Nantes - Hopital Laennec /ID# 212897, Saint-Herblain
- Orszagos Koranyi Pulmonologiai Intezet /ID# 213494, Budapest, Hungary
- Netherlands (2):
  - HagaZiekenhuis /ID# 212926, The Hague
  - Universitair Medisch Centrum Utrecht /ID# 212935, Utrecht
- New Zealand (4):
  - Greenlane Clinical Centre /ID# 221103, Epsom, Auckland
  - Christchurch Hospital /ID# 221105, Christchurch, Canterbury
  - Dunedin Hospital /ID# 221104, Otago, Otago
  - Waikato Hospital /ID# 221102, Hamilton, Waikato Region
- Szpital Dzieciecy Polanki /ID# 221330, Gdansk, Pomeranian Voivodeship, Poland
- Institut za zdravstvenu zastitu majke i deteta Srbije Dr Vukan Cupic /ID# 212820, Belgrade, Beograd, Serbia
- Slovakia (2):
  - Univerzitna nemocnica Bratislava Nemocnica Ruzinov /ID# 213146, Bratislava
  - Univerzitna nemocnica Bratislava Nemocnica Ruzinov /ID# 213596, Bratislava
- United Kingdom (8):
  - Barts Health NHS Trust /ID# 213016, London, London, City of
  - Nottingham University Hospitals NHS Trust /ID# 212531, Nottingham, Nottinghamshire
  - Cardiff & Vale University Health Board /ID# 212504, Cardiff, Wales
  - Royal Papworth Hospital NHS Foundation Trust /ID# 212507, Cambridge
  - Leeds Teaching Hospitals NHS Trust /ID# 212491, Leeds
  - Liverpool Heart and Chest Hospital NHS Foundation Trust /ID# 212291, Liverpool
  - Royal Brompton and Harefield Hospitals /ID# 212490, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 212665, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with Cystic Fibrosis (CF) who are homozygous for the F508del mutation were enrolled in this 2-part study to receive ABBV-3067 alone and in combination with ABBV-2222 for 28 days. In Part 1 participants received 2 different doses of ABBV-3067 as a single agent, and 5 different doses of ABBV-2222 as dual-combination therapy with ABBV-3067 at a fixed dose. Part 2 of the study was not conducted as it was deemed not enrollable by the time Part 1 was completed.
Period: Overall Study
Arm/Group | ABBV-3067 50 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + ABBV-2222 10 mg | ABBV-3067 150 mg + ABBV-2222 30 mg | ABBV-3067 150 mg + ABBV-2222 100 mg | ABBV-3067 150 mg + ABBV-2222 200 mg | ABBV-3067 150 mg + ABBV-2222 300 mg | Placebo for ABBV-3067 + Placebo for ABBV-2222
Started | 6 | 7 | 5 | 12 | 11 | 12 | 14 | 11
Completed | 6 | 7 | 4 | 12 | 11 | 12 | 13 | 10
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Not completed — Never Received Study Drug | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) includes all randomized participants who received at least 1 dose of study drug.
Groups:
- ABBV-3067 50 mg + Placebo for ABBV-2222: Participants received ABBV-3067 50 mg tablet orally QD plus placebo matching ABBV-2222 capsule, orally QD for 28 days.
- Total: Total of all reporting groups
Arm/Group | ABBV-3067 50 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + ABBV-2222 10 mg | ABBV-3067 150 mg + ABBV-2222 30 mg | ABBV-3067 150 mg + ABBV-2222 100 mg | ABBV-3067 150 mg + ABBV-2222 200 mg | ABBV-3067 150 mg + ABBV-2222 300 mg | Placebo for ABBV-3067 + Placebo for ABBV-2222 | Total
Number analyzed (Participants) | 6 | 7 | 5 | 12 | 11 | 12 | 14 | 11 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (4.46) | 31.6 (7.39) | 36.4 (15.50) | 33.8 (12.67) | 32.5 (12.53) | 32.5 (13.13) | 31.9 (9.00) | 26.8 (6.68) | 31.5 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 2 | 6 | 5 | 2 | 3 | 4 | 30
  Male | 1 | 4 | 3 | 6 | 6 | 10 | 11 | 7 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 7 | 5 | 12 | 11 | 12 | 14 | 11 | 78
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 7 | 5 | 12 | 11 | 12 | 14 | 11 | 78
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1 ) at Baseline [Mean (Standard Deviation); unit: percent predicted FEV1 (%)] — FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Population: Number analyzed are the number of participants with data available for analysis for ppFEV1 at baseline
  percent predicted FEV1 (%)
    number analyzed (Participants) | 6 | 7 | 4 | 12 | 11 | 12 | 13 | 11 | 76
    (all) | 67.0 (15.89) | 68.6 (11.16) | 65.8 (18.96) | 64.6 (16.84) | 68.1 (14.48) | 62.0 (15.18) | 67.6 (17.83) | 67.8 (13.19) | 66.3 (14.96)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline Through Day 29 in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration and is used as a measure of lung function. Mixed-effect model with repeated measures (MMRM) was used for the analyses.
Time Frame: Day 1 (Baseline) through Day 29
Population: FAS included all randomized participants who received at least 1 dose of study drug. Overall number of participants are the number of participants with data available for analyses.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted FEV1 (%)
Arm/Group | ABBV-3067 50 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + ABBV-2222 10 mg | ABBV-3067 150 mg + ABBV-2222 30 mg | ABBV-3067 150 mg + ABBV-2222 100 mg | ABBV-3067 150 mg + ABBV-2222 200 mg | ABBV-3067 150 mg + ABBV-2222 300 mg | Placebo for ABBV-3067 + Placebo for ABBV-2222
Number analyzed (Participants) | 5 | 5 | 2 | 5 | 10 | 11 | 11 | 9
percent predicted FEV1 (%) | 0.3 [-4.38 to 4.98] | -2.2 [-7.03 to 2.66] | 2.0 [-5.07 to 9.07] | 4.5 [-0.16 to 9.08] | 0.3 [-3.13 to 3.68] | 4.0 [0.79 to 7.28] | 2.4 [-0.85 to 5.74] | -2.2 [-5.83 to 1.43]

2. Secondary Outcome: Absolute Change From Baseline Through Day 29 in Sweat Chloride (SwCl)
Description: Sweat collection was performed to evaluate sweat chloride concentration. SwCl is a biomarker of cystic fibrosis transmembrane conductance regulator (CFTR) activity. Persons with CF have higher levels of chloride in their sweat. MMRM was used for the analysis.
Time Frame: Day 1 (Baseline) through Day 29
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | ABBV-3067 50 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + ABBV-2222 10 mg | ABBV-3067 150 mg + ABBV-2222 30 mg | ABBV-3067 150 mg + ABBV-2222 100 mg | ABBV-3067 150 mg + ABBV-2222 200 mg | ABBV-3067 150 mg + ABBV-2222 300 mg | Placebo for ABBV-3067 + Placebo for ABBV-2222
Number analyzed (Participants) | 5 | 7 | 3 | 11 | 10 | 12 | 13 | 9
millimole per liter (mmol/L) | -4.5 [-15.78 to 6.81] | -8.9 [-18.64 to 0.78] | -2.3 [-16.76 to 12.25] | -15.7 [-23.37 to -7.98] | -12.3 [-20.34 to -4.26] | -18.6 [-25.98 to -11.16] | -19.9 [-27.17 to -12.64] | -2.1 [-10.63 to 6.36]

3. Secondary Outcome: Absolute Change From Baseline Through Day 29 in Forced Vital Capacity (FVC)
Description: FVC is the total amount of air exhaled during forced expiratory volume (FEV) test and is a lung function test that is measured during spirometry. MMRM was used for the analyses.
Time Frame: Day 1 (Baseline) through Day 29
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: liter (L)
Arm/Group | ABBV-3067 50 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + ABBV-2222 10 mg | ABBV-3067 150 mg + ABBV-2222 30 mg | ABBV-3067 150 mg + ABBV-2222 100 mg | ABBV-3067 150 mg + ABBV-2222 200 mg | ABBV-3067 150 mg + ABBV-2222 300 mg | Placebo for ABBV-3067 + Placebo for ABBV-2222
Number analyzed (Participants) | 5 | 5 | 2 | 5 | 10 | 11 | 11 | 9
liter (L) | 0.0 [-0.22 to 0.23] | -0.0 [-0.24 to 0.20] | 0.0 [-0.28 to 0.35] | 0.1 [-0.16 to 0.28] | 0.1 [-0.08 to 0.24] | 0.0 [-0.11 to 0.19] | 0.0 [-0.12 to 0.19] | -0.2 [-0.38 to -0.03]

4. Secondary Outcome: Absolute Change From Baseline Through Day 29 in Forced Expiratory Flow at Mid-lung Capacity (FEF25-75)
Description: FEF25-75 is a lung function test that is measured during spirometry, and is defined as the forced expiratory flow between 25% and 75% of vital capacity (mid-lung capacity). MMRM was used for analyses.
Time Frame: Day 1 (Baseline) through Day 29
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: liter per seconds (L/sec)
Arm/Group | ABBV-3067 50 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + ABBV-2222 10 mg | ABBV-3067 150 mg + ABBV-2222 30 mg | ABBV-3067 150 mg + ABBV-2222 100 mg | ABBV-3067 150 mg + ABBV-2222 200 mg | ABBV-3067 150 mg + ABBV-2222 300 mg | Placebo for ABBV-3067 + Placebo for ABBV-2222
Number analyzed (Participants) | 5 | 5 | 2 | 5 | 10 | 11 | 11 | 9
liter per seconds (L/sec) | 0.0 [-0.27 to 0.29] | -0.0 [-0.29 to 0.27] | 0.2 [-0.26 to 0.57] | 0.2 [-0.08 to 0.47] | -0.0 [-0.23 to 0.18] | 0.3 [0.08 to 0.47] | 0.1 [-0.08 to 0.31] | 0.0 [-0.20 to 0.24]

5. Secondary Outcome: Relative Change From Baseline Through Day 29 in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration and is used as a measure of lung function. MMRM was used for analyses.
Time Frame: Day 1 (Baseline) through Day 29
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted FEV1
Arm/Group | ABBV-3067 50 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + ABBV-2222 10 mg | ABBV-3067 150 mg + ABBV-2222 30 mg | ABBV-3067 150 mg + ABBV-2222 100 mg | ABBV-3067 150 mg + ABBV-2222 200 mg | ABBV-3067 150 mg + ABBV-2222 300 mg | Placebo for ABBV-3067 + Placebo for ABBV-2222
Number analyzed (Participants) | 5 | 5 | 2 | 5 | 10 | 11 | 11 | 9
percent predicted FEV1 | 1.0 [-6.22 to 8.22] | -2.9 [-10.38 to 4.60] | 3.4 [-7.46 to 14.34] | 8.0 [0.87 to 15.14] | 1.4 [-3.82 to 6.69] | 5.7 [0.70 to 10.73] | 4.7 [-0.35 to 9.84] | -3.3 [-8.86 to 2.34]

6. Secondary Outcome: Relative Change From Baseline Through Day 29 in Forced Expiratory Flow at Mid-lung Capacity (FEF25-75)
Description: as for outcome 4
Time Frame: Day 1 (Baseline) through Day 29
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: L/sec
Arm/Group | ABBV-3067 50 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + ABBV-2222 10 mg | ABBV-3067 150 mg + ABBV-2222 30 mg | ABBV-3067 150 mg + ABBV-2222 100 mg | ABBV-3067 150 mg + ABBV-2222 200 mg | ABBV-3067 150 mg + ABBV-2222 300 mg | Placebo for ABBV-3067 + Placebo for ABBV-2222
Number analyzed (Participants) | 5 | 5 | 2 | 5 | 10 | 11 | 11 | 9
L/sec | 0.8 [-18.01 to 19.55] | -0.1 [-18.94 to 18.76] | 8.8 [-18.69 to 36.38] | 19.9 [1.61 to 38.28] | 0.1 [-13.46 to 13.65] | 18.5 [5.60 to 31.50] | 10.9 [-2.21 to 24.01] | 1.0 [-13.69 to 15.62]

7. Secondary Outcome: Relative Change From Baseline Through Day 29 in Forced Vital Capacity (FVC)
Description: FVC is the total amount of air exhaled during FEV test and is a lung function test that is measured during spirometry. MMRM was used for the analyses.
Time Frame: Day 1 (Baseline) through Day 29
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: liter
Arm/Group | ABBV-3067 50 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + ABBV-2222 10 mg | ABBV-3067 150 mg + ABBV-2222 30 mg | ABBV-3067 150 mg + ABBV-2222 100 mg | ABBV-3067 150 mg + ABBV-2222 200 mg | ABBV-3067 150 mg + ABBV-2222 300 mg | Placebo for ABBV-3067 + Placebo for ABBV-2222
Number analyzed (Participants) | 5 | 5 | 2 | 5 | 10 | 11 | 11 | 9
liter | 0.1 [-5.20 to 5.35] | -1.0 [-6.38 to 4.30] | 0.2 [-7.37 to 7.82] | 2.2 [-3.03 to 7.43] | 2.2 [-1.51 to 6.01] | 0.9 [-2.77 to 4.54] | 1.1 [-2.58 to 4.73] | -4.3 [-8.37 to -0.20]

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to end of study; maximum median time was 28.0 days. Treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) were collected from first dose of study drug until 30 days after last dose of study drug (Up to 63 days); mean duration on study drug was 28.3 days.
Description: All-cause mortality: all enrolled participants. SAEs and other adverse events: FAS includes all randomized participants who received at least 1 dose of study drug.
Arm/Group | ABBV-3067 50 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + Placebo for ABBV-2222 | ABBV-3067 150 mg + ABBV-2222 10 mg | ABBV-3067 150 mg + ABBV-2222 30 mg | ABBV-3067 150 mg + ABBV-2222 100 mg | ABBV-3067 150 mg + ABBV-2222 200 mg | ABBV-3067 150 mg + ABBV-2222 300 mg | Placebo for ABBV-3067 + Placebo for ABBV-2222
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/4 | 0/12 | 0/11 | 0/12 | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/4 | 2/12 | 0/11 | 0/12 | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 2/6 | 5/7 | 4/4 | 8/12 | 10/11 | 6/12 | 6/13 | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABBV-3067 50 mg + Placebo for ABBV-2222 (N=6) | ABBV-3067 150 mg + Placebo for ABBV-2222 (N=7) | ABBV-3067 150 mg + ABBV-2222 10 mg (N=4) | ABBV-3067 150 mg + ABBV-2222 30 mg (N=12) | ABBV-3067 150 mg + ABBV-2222 100 mg (N=11) | ABBV-3067 150 mg + ABBV-2222 200 mg (N=12) | ABBV-3067 150 mg + ABBV-2222 300 mg (N=13) | Placebo for ABBV-3067 + Placebo for ABBV-2222 (N=11)
ILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABBV-3067 50 mg + Placebo for ABBV-2222 (N=6) | ABBV-3067 150 mg + Placebo for ABBV-2222 (N=7) | ABBV-3067 150 mg + ABBV-2222 10 mg (N=4) | ABBV-3067 150 mg + ABBV-2222 30 mg (N=12) | ABBV-3067 150 mg + ABBV-2222 100 mg (N=11) | ABBV-3067 150 mg + ABBV-2222 200 mg (N=12) | ABBV-3067 150 mg + ABBV-2222 300 mg (N=13) | Placebo for ABBV-3067 + Placebo for ABBV-2222 (N=11)
CYSTIC FIBROSIS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYOPIA (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FAECES DISCOLOURED (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETCHING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACTERIURIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFECTIVE PULMONARY EXACERBATION OF CYSTIC FIBROSIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH PUSTULAR (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SIALOADENITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD GLUCOSE DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FORCED EXPIRATORY VOLUME DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
INCREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANIC ATTACK (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
INCREASED VISCOSITY OF UPPER RESPIRATORY SECRETION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PHARYNGEAL ERYTHEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RALES (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
SPUTUM INCREASED (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAPULE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT03969888/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/88/NCT03969888/SAP_001.pdf